CLINICAL TRIAL: NCT05381402
Title: COVID 19 Impact on Psoriasis Patients, a Hospital Based Study
Brief Title: Impact of COVID 19 on Psoriasis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, Dr, Cairo University
Other Study IDs: COVID 19 and psoriais patients
Record Dates: First submitted 2022-05-18; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: The Impact of COVID19 on Psoriasis Patients
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire to assess the impact of COVID 19 on psoriasis patients

SUMMARY:
The main objective of this work is to investigate the effect of COVID-19 pandemic on psoriasis patients.

This work is designed as a cross-sectional survey based on a questionnaire directed to Egyptian psoriasis patients.

ELIGIBILITY:
Inclusion Criteria:

* Psoriaisis patients

Exclusion Criteria:

* Children

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Psoriasis patients
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | 2-4 weeks
  To assess the effect of COVID 19 on psoriasis disease, treatment, follow up, vaccine